CLINICAL TRIAL: NCT01672645
Title: A Phase 1, Randomized, Double Blind, Placebo Controlled Study To Evaluate The Safety, Tolerability, Immunogenicity, And Exploratory Efficacy Of Multiple Ascending Dose Levels Of Pf-05402536 And Pf-06413367 In Healthy Adult Smokers
Brief Title: A Study to Assess the Safety and Tolerability of Different Doses of PF-05402536 and PF-06413367 in Healthy Adult Smokers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3771001
Record Dates: First submitted 2012-07-05; First posted 2012-08-27 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Smoking; Vaccines
Keywords: Smoking cessation; vaccine; Phase 1
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-05402536 (Experimental)
  Interventions: Biological: NIC7-001
- PF-06413367 (Experimental): Intramuscular, multiple dose
  Interventions: Biological: NIC7-003
- Placebo (Placebo Comparator): Intramuscular
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: NIC7-001 — Intramuscular, multiple dose
  Arms: PF-05402536
Biological: NIC7-003 — Intramuscular, multiple dose
  Arms: PF-06413367
Biological: Saline — Saline (0.9% sodium chloride)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability of multiple doses of PF-05402536 and PF-06413367 in healthy adult smokers.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smokers
* Males or females of non-child bearing potential, who are between the minimum legal age for smoking (approximately 18 or 19 years, depending on local jurisdiction) and 55 years, inclusive, and who are motivated to stop smoking.
* Subjects must have smoked an average of at least 10 cigarettes per day during the past year and during the month prior to the prescreening assessment for entry, with no period of abstinence greater than 3 months in the past year.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, or neurologic disease that may compromise their ability to safely participate in the study.
* Active suicidal ideation or history of suicidal behaviors within the past 5 years prior to the screening visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 277 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited local reactions (erythema, induration, and pain) and severity of the local reactions as self-reported on electronic diaries (e-diaries) for 7 days following vaccination. | Within 7 days after dose
Frequency of solicited systemic events (fever, vomiting, diarrhea, headache, fatigue, new or worsening muscle pain, and new or worsening joint pain) and severity of solicited systemic events as self-reported on e-diaries for 7 days following vaccination. | Within 7 days after dose
Number of Participants With Unsolicited Treatment-Emergent Adverse Events (AEs) by Seriousness and Relationship to Treatment | Baseline up to Day 364
Number of Participants With Abnormal Safety Laboratory Findings by Seriousness and Relationship to Treatment | Baseline up to Day 364

SECONDARY OUTCOMES:
Antibody titers against nicotine. | Up to Day 364
Avidity of antibodies against nicotine. | Up to Day 364
7-day point prevalence of smoking abstinence | Up to Day 364
4-week continuous abstinence rate from smoking | Up to Day 364
smoking behavioral measurements (including Minnesota Nicotine Withdrawal Scale, Modified Cigarette Evaluation Questionnaire, and Brief Questionnaire of Smoking Urges) | Up to Day 364

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Canada (3):
  - INC Research Toronto Inc., Toronto, Ontario
  - Diex Research Montreal, Inc., Montreal, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3771001&StudyName=A%20study%20to%20assess%20the%20safety%20and%20tolerability%20of%20different%20doses%20of%20PF-05402536%20and%20PF-06413367%20in%20healthy%20adult%20smokers.